CLINICAL TRIAL: NCT04296032
Title: Effects of Wearable Sensor Based Virtual Reality Game on Upper Extremity Function for Patients With Stroke
Brief Title: Effects of Virtual Reality Game on Upper Extremity Function for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB N201912049
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): Standard treatment 30 minutes plus virtual reality game 30 minutes, twice a week for 9 weeks.
  Interventions: Behavioral: virtual reality game traning; Behavioral: standard treatment
- standard treatment group (Active Comparator): Standard treatment 60 minutes, twice a week for 9 weeks.
  Interventions: Behavioral: standard treatment

INTERVENTIONS:
Behavioral: virtual reality game traning — The controllers were attached to upper extremity to control the game. The game could train the shoulder, elbow, and wrist control.
  Arms: virtual reality group
Behavioral: standard treatment — The program included bilateral hand, grasp/release, and pinch activities.

SUMMARY:
Virtual reality training had already been used in stroke rehabilitation, and previous studies supported that it could improve upper extremity ability and increase motivation and pleasure than conventional methods. Pablo is a new VR game combined with motion sensor system which can detect subject's activities. Unlike commercial camera systems such as Kinect or XBOX, the systems require a continuous sightline or enough active range of motion which may increase risk of compensatory movement. Few of studies had investigated the rehabilitation effects on upper extremity with Pablo for patients with stroke.The purpose of this study is to investigate the effects of virtual reality upper extremity training through Pablo system in patients with chronic stroke.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this study is to investigate the effects of virtual reality upper extremity training through Pablo system in patients with chronic stroke.

METHODS:Patients with mild to moderate motor deficits were recruited and randomly assigned to "VR plus standard rehabilitation group"(n=19), and "standard rehabilitation group" (n=19). After 12 training sessions (60 minutes a time, 2 times a week), the performance was assessed by a blinded assessor. The outcome measures included Fugl-Meyer Assessment-Upper Limb section(FMAUE), Box and block test(BBT), Dynanometer, active range of motion of shoulder and elbow,and Stroke Impact Scale.Modified Physical Activity Enjoyment Scale and adverse effect were recorded after each sessions.Collected data will be analyzed with sample T test by SPSS version 20.0, and alpha level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* First stroke with hemiplegia,
* Chronicity of >6 months
* Could understand instructions
* Brunnstrom stage of UE ≥IV.

Exclusion Criteria:

* Patients who were aged <20 years and >75 years
* Patients with visual or auditory impairment who were unable to see or hear the feedback from the device clearly
* Montreal Cognitive Assessment <16
* Modified Ashworth Scale score of >2
* Patients with other medical symptoms that can affect movement were excluded.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-upper extremity | Change from Baseline at 9 weeks
  The Fugl-Meyer Assessment-upper extremity (FMA-UE) measures motor impairment in the upper extremity. The assessment consists of 33 items, including movement, reflex, grasp, and coordination, and a total score of 66.

SECONDARY OUTCOMES:
Box and block test | Change from Baseline at 9 weeks
  The Box and block test (BBT) measures unilateral gross manual dexterity. The BBT score denotes the number of blocks transferred within 60 s.
Dynanometer | Change from Baseline at 9 weeks
  The grip dynamometer was used to measure the maximum isometric strength of the hand and forearm muscles. The mean score of 3 trials was calculated. For this measurement, the elbow was placed at 90° and the forearm was placed in mid-position.
Active range of motion of shoulder and elbow | Change from Baseline at 9 weeks
  The active range of motion of shoulder and elbow were measured through pablo system.
Stroke Impact Scale | Change from Baseline at 9 weeks
  The Stroke Impact Scale (SIS) is a quality of life measure designed specifically for patients with stroke. The instrument is a self-report questionnaire assessing eight domains: strength, hand function, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and social participation.
Modified Physical Activity Enjoyment Scale | Every training session during 18 sessions, total sessions continued to 9 weeks
  It is an scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7-point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it).
Adverse effect times | Every training session during 18 sessions, total sessions continued to 9 weeks
  To record the adverse effect times during the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hsinchieh Lee, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatano S. Experience from a multicentre stroke register: a preliminary report. Bull World Health Organ. 1976;54(5):541-53. PMID 1088404
- [Background] Carod-Artal J, Egido JA, Gonzalez JL, Varela de Seijas E. Quality of life among stroke survivors evaluated 1 year after stroke: experience of a stroke unit. Stroke. 2000 Dec;31(12):2995-3000. doi: 10.1161/01.str.31.12.2995. PMID 11108762
- [Background] Chiu L, Shyu WC, Liu YH. Comparisons of the cost-effectiveness among hospital chronic care, nursing home placement, home nursing care and family care for severe stroke patients. J Adv Nurs. 2001 Feb;33(3):380-6. doi: 10.1046/j.1365-2648.2001.01703.x. PMID 11251725
- [Background] Nordin N, Xie SQ, Wunsche B. Assessment of movement quality in robot- assisted upper limb rehabilitation after stroke: a review. J Neuroeng Rehabil. 2014 Sep 12;11:137. doi: 10.1186/1743-0003-11-137. PMID 25217124
- [Background] Jang SH. The recovery of walking in stroke patients: a review. Int J Rehabil Res. 2010 Dec;33(4):285-9. doi: 10.1097/MRR.0b013e32833f0500. PMID 20805757
- [Background] Kopp B, Kunkel A, Muhlnickel W, Villringer K, Taub E, Flor H. Plasticity in the motor system related to therapy-induced improvement of movement after stroke. Neuroreport. 1999 Mar 17;10(4):807-10. doi: 10.1097/00001756-199903170-00026. PMID 10208552
- [Background] Basteris A, Nijenhuis SM, Stienen AH, Buurke JH, Prange GB, Amirabdollahian F. Training modalities in robot-mediated upper limb rehabilitation in stroke: a framework for classification based on a systematic review. J Neuroeng Rehabil. 2014 Jul 10;11:111. doi: 10.1186/1743-0003-11-111. PMID 25012864
- [Background] Correction to: Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Dec;48(12):e369. doi: 10.1161/STR.0000000000000156. No abstract available. PMID 29180589
- [Background] Susanto EA, Tong RK, Ockenfeld C, Ho NS. Efficacy of robot-assisted fingers training in chronic stroke survivors: a pilot randomized-controlled trial. J Neuroeng Rehabil. 2015 Apr 25;12:42. doi: 10.1186/s12984-015-0033-5. PMID 25906983
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2015 Feb 12;2015(2):CD008349. doi: 10.1002/14651858.CD008349.pub3. PMID 25927099
- [Background] Smith, C., et al., Can non-immersive virtual reality improve physical outcomes of rehabilitation? Physical Therapy Reviews, 2012. 17(1): p. 1-15.
- [Background] Peters DM, McPherson AK, Fletcher B, McClenaghan BA, Fritz SL. Counting repetitions: an observational study of video game play in people with chronic poststroke hemiparesis. J Neurol Phys Ther. 2013 Sep;37(3):105-11. doi: 10.1097/NPT.0b013e31829ee9bc. PMID 23872681
- [Background] Laver, K.E., et al., Virtual reality for stroke rehabilitation. Stroke, 2018. 49(4): p. e160-e161.
- [Background] Lin LF, Lin YJ, Lin ZH, Chuang LY, Hsu WC, Lin YH. Feasibility and efficacy of wearable devices for upper limb rehabilitation in patients with chronic stroke: a randomized controlled pilot study. Eur J Phys Rehabil Med. 2018 Jun;54(3):388-396. doi: 10.23736/S1973-9087.17.04691-3. Epub 2017 Jun 19. PMID 28627862
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Derived] Kuo FL, Lee HC, Kuo TY, Wu YS, Lee YS, Lin JC, Huang SW. Effects of a wearable sensor-based virtual reality game on upper-extremity function in patients with stroke. Clin Biomech (Bristol). 2023 Apr;104:105944. doi: 10.1016/j.clinbiomech.2023.105944. Epub 2023 Mar 11. PMID 36963203